CLINICAL TRIAL: NCT00654134
Title: Inhalation of 20,000 EU of Clinical Center Reference Endotoxin in Healthy Volunteers
Brief Title: Inhalation of 20,000 Endotoxin Units(EU) of Clinical Center Reference Endotoxin in Healthy Volunteers
Acronym: Entox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Michelle Hernandez, MD, Assistant Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 05-2844 GCRC 2311; US EPA; NIEHS
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Clinical Center Reference Endotoxin — 20,000 EU inhaled

SUMMARY:
The purpose of this study is to determine the inflammatory response to 20,000 endotoxin units (EU) of CCRE (Clinical Center Reference Endotoxin) inhalation in a cohort of healthy volunteers. Preferably these subjects will have participated in ozone exposure studies, allowing a direct comparison of their responses to both endotoxin and ozone. Additionally, cardiovascular endpoints will be investigated with the CCRE exposure.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in Ozone Study
* Healthy adults
* Nonsmokers
* No chronic illness
* No active allergies

Exclusion Criteria:

* Reduced Lung function
* Asthma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To determine the inflammatory response to 20,000 endotoxin units (EU) of CCRE (Clinical Center Reference Endotoxin) inhalation in a cohort of healthy volunteers. | 6 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina
Locations (1):
- Us Epa Hsf, Chapel Hill, North Carolina, United States